CLINICAL TRIAL: NCT04661904
Title: Effect of Continuous Theta Burst Stimulation (cTBS) on Postoperative Delirium
Brief Title: Continuous Theta Burst Stimulation (cTBS) and Postoperative Delirium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yuan Shen, MD, PhD, Chief of Psychiatry, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: dsyy005
Record Dates: First submitted 2020-11-26; First posted 2020-12-10 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Delirium; Transcranial Magnetic Stimulation, Repetitive
Keywords: postoperative delirium; continuous theta burst stimulation
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cTBS group (Experimental): Patients randomly assigned to cTBS group received 9 sessions cTBS for total three days after surgery.
  Interventions: Device: Continuous theta burst stimulation (cTBS)
- sham group (Sham Comparator): Patients randomly assigned to sham group received 9 sessions sham stimulation for total three days after surgery.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Continuous theta burst stimulation (cTBS) — Our active treatment consisted of 600 pulses per session, delivered over the right dorsolateral prefrontal cortex at 80% of resting motor threshold (RMT). Every session cTBS consists of 50 Hz triplets of pulses delivered at 5 Hz for 40 seconds for a total of 600 pulses. Every set simulation includes 3 sessions. All enrolled patient in the cTBS group received 1 set simulation per day with an intersession interval (ISI) of over 30 minutes during the hospitalization after the surgery. The first set of stimulation was given at 4 hours after the end of surgery on the day of surgery. The other sets of stimulation were given at 8 am, 8:30 am and 9:00 am on postoperative day 1and 2, respectively.
  Arms: cTBS group
Device: Sham stimulation — The sham stimulation group received a sham cTBS (600 pulses per session, 3 sessions per day, ISI ≥ 30mins, 3 days) with the coil set at 90 against the skull. The first set of stimulation was given at 4 hours after the end of surgery on the day of surgery. The other sets of stimulation were given at 8 am, 8:30 am and 9:00 am on postoperative day 1 and 2, respectively.
  Arms: sham group

SUMMARY:
To investigate the impact of cTBS on the incidence of postoperative delirium and changes of cognitive function in elderly patients after surgery. To explore whether short-term cTBS can reduce the risk of postoperative delirium as a preventive strategy.

DETAILED DESCRIPTION:
Postoperative delirium is the most common postoperative complications among elderly. Nevertheless, there remains no effective medication or intervention been approved in postoperative delirium. Recent research suggests that continuous theta burst stimulation (cTBS) has shown positive effect on improving global cognitive function in multiple mental disorders. However, the effects on cognitive function in postoperative delirium remain uninvestigated.

ELIGIBILITY:
Participants were included if they:

1. were 65 years old or older;
2. had orthopedic surgery under general anesthesia;
3. had normal cognitive function at enrolment [for illiterate, Mini-Mental State Examination (MMSE) ≥ 17; for individuals with 1-6 years of education, MMSE ≥ 20; for individuals with 7 or more years of education, MMSE ≥ 24];
4. were able to complete cognitive assessments and the Confusion Assessment Method (CAM);
5. Chinese Mandarin as their native language;
6. were willing to participate and being competent to provide informed consent.

Patients were excluded if they:

1. had delirium assessed by CAM before surgery;
2. had neurological diseases (e.g., stroke, Parkinson's disease, etc.) according to International Statistical Classification of Diseases and Related Health Problems 11th Revision (ICD-11);
3. had mental disorders (e.g., major depressive disorder, dementia, etc.) according to Diagnostic and Statistical Manual of Mental Disorders (Fifth Edition) (DSM-5);
4. had contraindications of cTBS (e.g., head trauma, history of epilepsy or metal implants in the head);
5. participating in other clinical studies at the time of screening;
6. having postoperative complications such as pulmonary infection, pulmonary embolism and stroke.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 324 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | 3 days after surgery
  Incidence of postoperative delirium on postoperative day 1, 2 and 3 was defined according to the confusion assessment methods (CAM).
Cognitive function related to delirium | 3 days after surgery
  The cognitive function related to delirium was assessed by using Delirium Symptom Interview Daily (DSI Daily).
Severity of postoperative delirium | 3 days after surgery
  Severity of postoperative delirium on postoperative day 1, 2 and 3 was defined according to he Confusion Assessment Method based delirium severity evaluation tool (CAM-S).The sum score of CAM-S ranges from 0 (no) to 19 (most severe).

SECONDARY OUTCOMES:
Pain level | 3 days after surgery
  This was assessed by using Visual Analogue Scale (VAS). The patients scored according to the severity of their pain from no pain (0) to most painful (10).
Sleep quality | 3 days after surgery
  leep Quality was assessed by the Pittsburgh Sleep Quality Index (PSQI) at baseline (T0), and DSI Daily after surgery.The global PSQI score ranges from 0 to 21, where lower scores denote a healthier sleep quality.
Ability of daily living | up to 7 days after anesthesia/surgery
  This was assessed by using Chinese version of Activity of Daily Living (ADL) Scale.The total score of ADLs ranges from 14 to 56 points and higher ADLs scores indicate lower activities of daily living.
Rate of complication and mortality | up to 7 days after anesthesia/surgery
  Rate of complication and mortality during the stay in hospital or up to 7 days after anesthesia/surgery, depending which one is longer

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Shen, MD, PhD, Principal Investigator — Shanghai, Shanghai, China, 200072
Locations (1):
- Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wei X, Wang M, Ma X, Tang T, Shi J, Zhao D, Yuan T, Xie Z, Shen Y. Treatment of postoperative delirium with continuous theta burst stimulation: study protocol for a randomised controlled trial. BMJ Open. 2021 Aug 16;11(8):e048093. doi: 10.1136/bmjopen-2020-048093. PMID 34400453